CLINICAL TRIAL: NCT05640518
Title: External Validation of the VExUS Score for the Prediction of Acute Renal Failure in Cardiac Surgery
Acronym: ValiVexus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0274
Record Dates: First submitted 2022-10-20; First posted 2022-12-07 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-10

CONDITIONS: Renal Failure; Acute Renal Failure; Renal Insufficiency; Acute Renal Insufficiency
Keywords: Renal failure; Cardiac surgery; VExUS score; venous congestion
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute renal failure is a frequent complication associated with significant morbidity and mortality in postoperative cardiac surgery.

The VExUS (Venous Excess UltraSound grading system) score was created to qualitatively assess this venous congestion, based on ultrasound data from patients obtained post operatively in cardiac surgery. These data included: inferior vena cava diameter, Doppler flow of the suprahepatic veins, portal trunk and renal veins.

This score is predictive of the onset of acute renal failure in the first 3 days after surgery.

The VExUS score has not been validated in an external and prospective way in cardiac surgery.

DETAILED DESCRIPTION:
Acute renal failure is a frequent complication associated with significant morbidity and mortality in postoperative cardiac surgery.

The pathophysiology in this context is complex, poorly understood and the causes are multiple: underlying nephropathy, intra- or postoperative haemodynamic instability, the use of an extracorporeal circulation, inflammation, etc.

One of the other possible etiologies is venous congestion. This may be due to volume overload and/or isolated global or right heart dysfunction.

Early treatment could prevent the onset of ARF or reduce its consequences, hence the importance of being able to predict its onset.

The VExUS (Venous Excess UltraSound grading system) score was created to qualitatively assess this venous congestion, based on ultrasound data from patients obtained post operatively in cardiac surgery. These data included: inferior vena cava diameter, Doppler flow of the suprahepatic veins, portal trunk and renal veins.

This score is predictive of the onset of acute renal failure in the first 3 days after surgery.

The VExUS score has not been validated in an external and prospective way in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled cardiac surgery
* Affiliated to a social security system

Exclusion Criteria:

* Emergency surgery
* Chronic renal failure defined by a glomerular filtration rate of less than 30ml/min or dialysis.
* renal transplant recipients
* Cirrhosis and portal hypertension
* Setting up a left ventricular assist device implantation
* Patient under ECMO (ExtraCorporeal Membrane Oxygenation), intra-aortic balloon pump, or a mechanical circulatory support device such as IMPELLA
* No available operator to perform ultrasound scans
* Patients objecting to the use of their data in research
* Subject under guardianship or subject deprived of freedom
* Pregnant or breastfeeding women
* Resume surgery within 48 hours of scheduled surgery
* Lack of a trained operator to perform D+1 and D+2 ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for cardiac surgery will be screened. They will be referred to the preoperative anesthesia consultation by the cardiac surgeons, which is a legal requirement in France.
  The geographical area of origin corresponds to the recruitment area of the cardiac surgery department of the Grenoble-Alpes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Association between the change in ultrasound data collected in the VExUS score and postoperative acute renal failure (defined by a creatininemia increase by 26.5 µmol/L in 48 hours). | From date of randomization until date of post-operative acute renal failure (detected by daily creatininemia), assessed up to a variable period of time estimated to 2 weeks.
  correlation between operator in term of VExUS staging (VExUS score will be assessed at day 1, 2 and 3 after the surgery, in intensive care unit.
Association between the change in ultrasound data collected in the VExUS score and postoperative acute renal failure. | From date of randomization until date of post-operative acute renal failure (detected by daily creatininemia), assessed up to a variable period of time estimated to 2 weeks
  Specificity of the VExUS score to predict an acute kidney failure will be evaluated

SECONDARY OUTCOMES:
Correlation between the VExUS score and a postoperative acute renal failure | 3 days
  Use of a multivariable COX regression to evaluate the correlation between the VExUS score measured at day 1, 2 and 3 and a post-operative acute renal failure during the stay in intensive care unit
Diagnostic performances of the VExUS Score for postoperative acute renal failure | 3 days
  Sensitivity, NPV, PPV
Correlation between central venous pressure (CVP) and postoperative acute renal failure. If a statistical association is present, diagnostic performance (Sensitivity, Specificity, NPV, PPV) of the value | 3 days
  Central venous pressure (CVP). The values will be taken during the ultrasound scans at Day 0, Day 1 and Day 2. The units of pressure are mmHg. A value greater than 12mmHg will be considered high, a lower value as not high. The CVP is measured by a central venous line.
Correlation between daily fluid balance and postoperative acute renal failure. If a statistical association is present, diagnostic performance (Sensitivity, Specificity, NPV, PPV) of the value | 3 days
  Water balance: 24-hour input-output balance, in millilitres, collected daily. Values measured at Day 0, Day 1, Day 2
Correlation between daily fluid balance and postoperative acute renal failure. If a statistical association is present, diagnostic performance (Sensitivity, Specificity, NPV, PPV) of the value | 3 days
  Water balance: including the weight in Kg compared to the reference weight established during the anaesthetic consultation. Values measured at Day 0, Day 1, Day 2
Correlation between an isolated component of the VExUS score, echocardiography and postoperative acute renal failure. If a statistical association is present, diagnostic performance (Sensitivity, Specificity, NPV, PPV) of the value | 3 days
  An isolated component of the VExUS score that is measured at D0; D1; D2 by ultrasound
  1. Inferior vena cava diameter
  2. Doppler profile of the suprahepatic vein
  3. Doppler profile of portal vein
  4. Renal vein Doppler profile
Correlation between an echocardiographic abnormality and postoperative acute renal failure. If a statistical association is present, diagnostic performance (Sensitivity, Specificity, NPV, PPV) of the value. | 3 days
  Ultrasound assessment of the left and right heart: Visual LVEF, sub-aortic LTI, Mitral Doppler (E wave, A wave, E/A ratio, deceleration time), LV/VD ratio (less than or greater than 0.6); TAPSE (unit: mm); S wave (unit: cm/seconds); LTI flow (unit: m/seconds); diameter (unit: mm) and ICV compliance. Values also taken at D0, D1 and D2.
Correlation between VExUS score and the use of extra renal replacement therapy | From randomization until date of postoperative need of extra renal replacement therapy, assessed up to a variable period of time estimated to 2 weeks.
  Use of extra renal replacement therapy: based on dialysis prescriptions, binary value (yes/no) regardless of the method used (CVVHF, CVVHDF, CVVHD)
Correlation between VExUS score and length of stay | From randomization until date of discharge, assessed up to a variable period of time estimated to 2 weeks.
  Length of stay in days: in intensive care, cardiac surgery and rehabilitation. Determined thanks to medical records.
Correlation between VExUS score and 1-month mortality | 1 month after admission in intensive care
  Mortality: binary (yes/no) at 1 month. The data will be collected by phone call to the patient or a relative, or by consulting the medical record.
Correlation between renal arterial resistance index and postoperative acute renal failure. If a statistical association is present, diagnostic performance (Sensitivity, Specificity, NPV, PPV) | 3 days
  Renal arterial resistance index are measured at D0; D1; D2 during the ultrasound scans.
Correlation between renal venous impedance index and postoperative acute renal failure. If a statistical association is present, diagnostic performance (Sensitivity, Specificity, NPV, PPV) | 3 days
  Veinous impedance index are measured at D0; D1; D2 during the ultrasound scans.

CONTACTS AND LOCATIONS:
Overall Officials: Timothée ABAZIOU, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoste EA, Cruz DN, Davenport A, Mehta RL, Piccinni P, Tetta C, Viscovo G, Ronco C. The epidemiology of cardiac surgery-associated acute kidney injury. Int J Artif Organs. 2008 Feb;31(2):158-65. doi: 10.1177/039139880803100209. PMID 18311732
- [Background] Beaubien-Souligny W, Benkreira A, Robillard P, Bouabdallaoui N, Chasse M, Desjardins G, Lamarche Y, White M, Bouchard J, Denault A. Alterations in Portal Vein Flow and Intrarenal Venous Flow Are Associated With Acute Kidney Injury After Cardiac Surgery: A Prospective Observational Cohort Study. J Am Heart Assoc. 2018 Oct 2;7(19):e009961. doi: 10.1161/JAHA.118.009961. PMID 30371304
- [Background] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297
- [Background] Bossard G, Bourgoin P, Corbeau JJ, Huntzinger J, Beydon L. Early detection of postoperative acute kidney injury by Doppler renal resistive index in cardiac surgery with cardiopulmonary bypass. Br J Anaesth. 2011 Dec;107(6):891-8. doi: 10.1093/bja/aer289. Epub 2011 Sep 22. PMID 21940396